CLINICAL TRIAL: NCT04693208
Title: Analgesic Effect of Laser Therapy in Paediatric Patients Undergoing Tonsillectomy
Brief Title: Analgesic Effect of Laser Therapy in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adverse reactions (tonsillar bleeding after treatment)
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC 02/2020
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative
Keywords: Pain; Tonsillectomy; Laser Therapy; Photo-biomodulation
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): Laser light will be applied to the surgery site after tonsils excision.
  Interventions: Device: Laser therapy
- Standard care (No Intervention)

INTERVENTIONS:
Device: Laser therapy — Laser treatment parameters will be two combined wavelength (660 and 970 nm), 3.2 Watt peak power, 320 milliWatt/cm2, 36.8 Joule/cm2 fluency, and 50% frequency, for a total time of 3 minutes for each site
  Arms: Laser

SUMMARY:
Pain management after tonsillectomy could be challenging, with different protocols and various outcome depending on individual patient; moreover, odynophagia due to surgery can, in extreme cases, lead to block oral fluid intake, ending in dehydration and thus hospitalization. A small pilot study demonstrated efficacy of photo-biomodulation (PBM) in managing pain after tonsillectomy and it suggests that PBM can be included in clinical practice. The present research aims to confirm and expand the findings from this study, being the first step in including PBM in clinical routine after tonsillectomy. Use of this treatment, which is non-damaging, non-toxic and easy to supply to patients, could greatly improve individual quality of life after a surgical treatment; its use in the clinical practice could represent an advantage for the institute, leading to more patients' satisfaction, due to the lower pain sensation after surgery and quicker recovery time.

ELIGIBILITY:
Inclusion Criteria:

Tonsillectomy or adenotonsillectomy due to apneic chronic snoring and/or obstructive sleep apnea and/or recurrent tonsillitis

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) Score > 2
2. Neuropsychiatric co-morbidity
3. Pro-hemorrhage coagulation disorders

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Reduction in pain score, age 3-7 years | After 24 hours
  The score is evaluated using the Wong-Baker scale, ranged 0-10. Higher scores correspond to higher levels of pain.
Reduction in pain score, age 8-18 years | After 24 hours
  The score is evaluated using a Visual Analogue Scale (VAS) ranged 0-10. Higher scores correspond to higher levels of pain.

SECONDARY OUTCOMES:
Reduction in pain score, age 3-7 years | After 4 hours
  The score is evaluated using the Wong-Baker scale, ranged 0-10. Higher scores correspond to higher levels of pain.depending on age
Reduction in pain score, age 3-7 years | After 6 hours
  The score is evaluated using the Wong-Baker scale, ranged 0-10. Higher scores correspond to higher levels of pain.
Reduction in pain score, age 8-18 years | After 4 hours
  The score is evaluated using a Visual Analogue Scale (VAS) ranged 0-10. Higher scores correspond to higher levels of pain.
Reduction in pain score, age 8-18 years | After 6 hours
  The score is evaluated using a Visual Analogue Scale (VAS) ranged 0-10. Higher scores correspond to higher levels of pain.
Frequency of use of pain killer drugs | Within 24 hours
  Number of postoperative pain killers drugs administered
Reduction in pain score evaluated by parents | 7 days after discharge
  Pain evaluated by parents using a Visual Analogue Scale (VAS) ranged 0-10. Higher scores correspond to higher levels of pain.
Quality of sleep | 7 days after discharge
  The quality of children sleep will be evaluated by parents or caregivers through a questionnaire
Mean daily food intake. | 7 days after discharge
  The mean daily food intake of children will be evaluated by parents or caregivers through a questionnaire.
Frequency of use of pain killer drugs | 7 days after discharge
  The number of pain killers drugs administered at home will be measured by parents or caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Sagredini, MD, Study Chair — Institute for Maternal and Child Health IRCCS Burlo Garofolo; Eva Orzan, MD, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste, Italy